CLINICAL TRIAL: NCT04218084
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Voxelotor (GBT440) in Pediatric Participants With Sickle Cell Disease (HOPE Kids 2)
Brief Title: Study to Evaluate the Effect of GBT440 on TCD in Pediatrics With Sickle Cell Disease
Acronym: HOPE Kids 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Emerging clinical data evaluated by Pfizer and shared with regulatory authorities indicates that the risk profile of voxelotor in people with SCD exceeds the benefits observed in previously generated global research and requires further assessment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBT440-032; 2017-000903-26 (EudraCT Number); C5341021 (Other: Alias Study Number)
Expanded Access: NCT04724421 (No longer available)
Record Dates: First submitted 2019-12-20; First posted 2020-01-06 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Transcranial Doppler Ultrasound (TCD)
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind, Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Voxelotor (Experimental): Voxelotor 1500mg or equivalent daily as a tablet, dispersible tablet, or as powder for oral suspension.
  Interventions: Drug: Voxelotor
- Placebo (Placebo Comparator): Matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Voxelotor — Participants are randomized 1:1 to receive voxelotor or placebo.
  Arms: Voxelotor
Drug: Placebo — Matching placebo.
  Arms: Placebo

SUMMARY:
This study is a Phase 3, randomized, double-blind, placebo-controlled study of voxelotor in pediatric participants, aged ≥ 2 to < 15 years old, with Sickle Cell Disease. The primary objective is to evaluate the effect of voxelotor on the TCD (Transcranial Doppler Ultrasound) measurements in SCD participants in this age range.

DETAILED DESCRIPTION:
This study is a Phase 3, randomized, double-blind, placebo-controlled study of voxelotor in pediatric participants, aged ≥ 2 to < 15 years old, with Sickle Cell Disease. The study will be conducted at approximately 50 international clinical sites, and will enroll approximately 224 participants. Participants will be randomized in a 1:1 ratio to receive voxelotor or placebo. All participants younger than 12 years of age and randomized to voxelotor will receive a dose based on their body weight, to provide exposure corresponding to the adult dose of 1500 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with Sickle Cell Anemia (SCA) HbSS, HbSβ0 thalassemia genotype
2. TCD time averaged maximum of the mean velocity (TAMMV) arterial cerebral blood flow ≥ 170 to < 200cm/sec during the Screening Period
3. Hb ≥ 5.5 and ≤ 10.5 g/dL during screening
4. For participants taking HU, the dose of HU (mg/kg) must be stable for at least 90 days prior to signing the informed consent form (ICF) and/or assent form, and with no anticipated need for dose adjustments (other than weight based) or for initiation of HU for non-chronic use during the study, in the opinion of the Investigator
5. Written informed parental/guardian consent and participant assent (where applicable) has been obtained per IRB/EC policy and requirements, consistent with ICH guidelines.

Exclusion Criteria:

1. Body weight < 10kg at the screening visit
2. Hospitalization for VOC or acute chest syndrome (ACS) within the 14 days prior to execution of informed consent/assent
3. More than 10 VOCs within the past 12 months that required hospitalization, emergency room, or clinic visit
4. Stroke resulting in focal neurological deficit; previous silent infarcts are permitted.
5. Known history or findings suggestive of significant cerebral vasculopathy
6. History of seizure disorder
7. Has been treated with erythropoietin or other hematopoietic growth factors within 28 days of signing informed consent/assent or if, in the opinion of the Investigator, there is an anticipated need for such agents during the study
8. RBC transfusion therapy (also termed chronic, prophylactic, or preventative transfusion) or has received an RBC transfusion or exchange transfusion for any reason within 90 days of signing the informed consent/assent

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (8):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta: Hughes Spalding, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Hospital- Wallace Tower, Houston, Texas
- Egypt (4):
  - Alexandria Clinical Research Center, Faculty of Medicine, Alexandria University, Alexandria
  - Zagazig University Hospital, Alexandria
  - Abu El Rich Hospital, Cairo University Hospital, Cairo
  - Ain Shams University Hospital-Clinical Research Center (MASRI), Cairo
- Ghana (2):
  - Department of Child Health, University of Ghana Medical School, College of Health Sciences, Accra
  - Komfo Anokye Teaching Hospital, Kumasi
- Italy (3):
  - Azienda Ospedaliera Universitaria (AOU) Meyer, Florence
  - Azienda Ospedaliera Universitaria (A.O.U.) "Luigi Vanvitelli", Napoli
  - Azienda Ospedaliera Universita (AOU) Padova, Padua
- Kenya (4):
  - Kemri/Crdr,Siaya,Kemri Clinical Research Annex, Kisumu, Siaya County
  - KEMRI CRDR Clinical Research Annex, Nairobi
  - Strathmore University Medical Centre, Nairobi
  - Gertrude's Children Hospital, Nairobi
- Nigeria (5):
  - University of Nigeria Teaching Hospital, Enugu
  - College of Medicine, University of Ibadan, Ibadan
  - Barau Dikko Teaching/ Kaduna State University, Kaduna
  - Aminu Kano Teaching Hospital, Kano
  - Lagos University Teaching Hospital, Lagos
- Sultan Qaboos University Hospital, Muscat, Oman
- King Abdullah International Medical Research Center (KAIMR) Ministry of National Guard - Health, Riyadh, Saudi Arabia
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-032

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 236 participants were assigned to the study treatment. Results are presented for only primary outcome measure. Remaining outcome measures would be reported upon completion of their analysis at study completion date. Data cut-off date for this study was 18-Jan-2024.
Groups:
- Voxelotor: Participants aged greater than or equal to 12 years of age received 1500 milligrams (mg) voxelotor tablet orally once daily for 96 weeks. Participants less than 12 years of age received voxelotor at a weight based (1500 mg-equivalent) dose. Participants were followed up to 4 weeks after last dose of study drug.
- Placebo: Participants received voxelotor matched placebo orally once daily for 96 weeks. Participants were followed up to 4 weeks after last dose of study drug.
Period: Overall Study
Arm/Group | Voxelotor | Placebo
Started | 120 | 116
Completed | 25 | 23
Not Completed | 95 | 93
Not completed — Adverse Event | 7 | 2
Not completed — Withdrawal of Consent | 4 | 5
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Non-compliance with study drug | 1 | 1
Not completed — Abnormal transcranial doppler (TCD) | 19 | 24
Not completed — Other | 0 | 1
Not completed — Ongoing at data cut-off date | 62 | 58

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Voxelotor: Participants aged greater than or equal to 12 years of age received 1500 mg voxelotor tablet orally once daily for 96 weeks. Participants less than 12 years of age received voxelotor at a weight based (1500 mg-equivalent) dose. Participants were followed up to 4 weeks after last dose of study drug.
- Total: Total of all reporting groups
Arm/Group | Voxelotor | Placebo | Total
Number analyzed (Participants) | 120 | 116 | 236
Age, Customized [Count of Participants; unit: Participants]
  Age: 2 to less than (<) 4 Years | 14 | 10 | 24
  Age: 4 to < 12 Years | 91 | 92 | 183
  Age: 12 to < 15 Years | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 63 | 59 | 122
  Sex: Male | 57 | 57 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 0 | 1
  Ethnicity: Not Hispanic or Latino | 114 | 113 | 227
  Ethnicity: Unknown or Not Reported | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was reported.
  Participants
    Race: African | 69 | 80 | 149
    Race: Arab | 12 | 11 | 23
    Race: Black or African American | 8 | 2 | 10
    Race: White | 2 | 0 | 2
    Race: Multi-Racial | 29 | 23 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time-Averaged Maximum of Mean Velocity (TAMMV) Arterial Cerebral Blood Flow at Week 24
Description: TAMMV was defined as the time averaged maximum of the mean velocity arterial cerebral blood flow and was measured using transcranial Doppler (TCD). Analysis was performed using mixed model for repeated measures (MMRM) including treatment, study visit, treatment by visit interaction, baseline hydroxyurea (HU) use (yes; no), age group (2 to <= 8 years; >8 to <15 years), and baseline TAMMV value (170 centimeter per second [cm/sec] to < 185 cm/sec; 185 cm/sec to < 200 cm/sec) as fixed effect terms and used a compound symmetry covariance matrix for within-participant variability.
Time Frame: Baseline (value at screening), Week 24
Population: ITT analysis population included all randomized participants. Here, "Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeter per second (cm/sec)
Groups:
- Voxelotor: Participants aged 12 years or older were received 1500 milligrams (mg) voxelotor orally once daily for 96 weeks. Participants aged 2 to less than 12 years of age received voxelotor at a weight based (1500 mg-equivalent) dose.
- Placebo: Participants received voxelotor matched placebo orally once daily for 96 weeks.
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 108 | 114
Centimeter per second (cm/sec) | -12.15 [-15.83 to -8.46] | -4.42 [-8.23 to -0.61]
Statistical Analysis 1: Comparison: Voxelotor vs Placebo; Week 24; Test type: Other — Mixed Model Repeated Measures analysis; p = 0.0043, Mixed Models for Repeated Measures; Difference in LS mean = -7.73, 95% CI 2-sided [-13.03 to -2.42]

2. Secondary Outcome: Change From Baseline in Transcranial Doppler (TCD) Flow Velocity at Week 48.
Description: Change in TCD flow velocity from baseline to week 48 was analyzed using the MMRM model including treatment, study visit, treatment by visit interaction, baseline hydroxyurea use (yes; no), age group (2 to <= 8 years; >8 to <15 years), and baseline TAMMV value (170 cm/sec to < 185 cm/sec; 185 cm/sec to < 200 cm/sec) as fixed effect terms and used a compound symmetry covariance matrix for within-subject variability.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

3. Secondary Outcome: Time to Conversion to Abnormal TCD Flow
Description: Time to conversion was the number of weeks from the date of randomization to the date of TCD assessment when an abnormal TCD flow velocity (>= 200 cm/sec) is determined.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

4. Secondary Outcome: Time to Reversion to Normal TCD Flow
Description: Time to first normal TCD flow was the number of weeks from randomization to the date of first normal (<170 cm/sec) TCD flow.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

5. Secondary Outcome: Percentage of Participants With TCD Flow Velocity Reduction Greater Than or Equal to (>=)15 cm/Sec at Weeks 24 and 48
Description: TCD flow velocity reduction from Baseline ≥ 15 cm/sec at week 24, week 48 was analyzed using an exact Cochran-Mantel-Haenszel (CMH) general association test stratified for baseline HU use (yes; no), age group (2 to <= 8 years; >8 to <15 years), and baseline TAMMV value (170 cm/sec to < 185 cm/sec; 185 cm/sec to < 200 cm/sec).
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

6. Secondary Outcome: Change From Baseline in Hemoglobin (Hb) at Weeks 24 and 48
Description: Change from baseline in hemoglobin at weeks 24 and 48 was analyzed using the MMRM model including treatment, study visit, treatment by visit interaction, baseline hydroxyurea use (yes; no), age group (2 to <= 8 years; >8 to <15 years) and baseline TAMMV value (170 centimeter per second [cm/sec] to < 185 cm/sec; 185 cm/sec to < 200 cm/sec) as fixed effect terms and used a compound symmetry covariance matrix for within-participant variability.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

7. Secondary Outcome: Percent Change From Baseline in Unconjugated Bilirubin at Weeks 24 and 48
Description: Percent change from baseline in unconjugated bilirubin at weeks 24 and 48 was reported in this outcome measure. Analysis was performed using MMRM including treatment, study visit, treatment by visit interaction, baseline hydroxyurea use (yes; no), age group (2 to <= 8 years; >8 to <15 years), and baseline TAMMV value (170 centimeter per second [cm/sec] to < 185 cm/sec; 185 cm/sec to < 200 cm/sec) as fixed effect terms and used a compound symmetry covariance matrix for within-subject variability.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

8. Secondary Outcome: Percent Change From Baseline in Reticulocyte at Weeks 24 and 48
Description: Percent change from baseline in reticulocyte at weeks 24 and 48 was reported in this outcome measure. Analysis was performed using MMRM including treatment, study visit, treatment by visit interaction, baseline hydroxyurea use (yes; no), age group (2 to <= 8 years; >8 to <15 years), and baseline TAMMV value (170 centimeter per second [cm/sec] to < 185 cm/sec; 185 cm/sec to < 200 cm/sec) as fixed effect terms and used a compound symmetry covariance matrix for within-participant variability.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

9. Secondary Outcome: Percent Change From Baseline in Absolute Reticulocyte at Weeks 24 and 48
Description: Percent change from baseline in absolute reticulocyte at weeks 24 and 48 was reported in this outcome measure. Analysis was performed using MMRM including treatment, study visit, treatment by visit interaction, baseline hydroxyurea use (yes; no), age group (2 to <= 8 years; >8 to <15 years), and baseline TAMMV value (170 centimeter per second [cm/sec] to < 185 cm/sec; 185 cm/sec to < 200 cm/sec) as fixed effect terms and used a compound symmetry covariance matrix for within-subject variability.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

10. Secondary Outcome: Percent Change From Baseline in Lactate Dehydrogenase (LDH) at Weeks 24 and 48
Description: Percent change from baseline in LDH at weeks 24 and 48 was reported in this outcome measure. Analysis was performed using MMRM including treatment, study visit, treatment by visit interaction, baseline hydroxyurea use (yes; no), age group (2 to <= 8 years; >8 to <15 years), and baseline TAMMV value (170 centimeter per second [cm/sec] to < 185 cm/sec; 185 cm/sec to < 200 cm/sec) as fixed effect terms and used a compound symmetry covariance matrix for within-subject variability.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

11. Secondary Outcome: Annualized Incidence Rate of Vaso-Occlusive Crises (VOCs)
Description: VOC was defined as a composite of acute painful crisis and/or acute chest syndrome (ACS). Annualized incidence rate was defined as total number of events per total person-years. Total person-years was the sum of participants treatment period in years, which included the time from randomization date to the earliest of (last dose date, post-randomization initiation for participants with no hydroxyurea at baseline, end of study, and data cutoff date). The 95% CI of rate displayed the exact Poisson confidence limits.
Time Frame: From treatment initiation till study completion
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: From Day 1 up to 28 days after last dose of study drug (maximum treatment exposure was 106 weeks)
Description: Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Voxelotor | Placebo
All-Cause Mortality (participants affected / at risk) | 6/120 | 2/116
Serious Adverse Events (participants affected / at risk) | 48/120 | 24/116
Other Adverse Events (participants affected / at risk) | 40/120 | 27/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voxelotor (N=120) | Placebo (N=116)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 42 | 19
Anaemia (Blood and lymphatic system disorders) | 10 | 9
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 2
Pneumonia viral (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 18 | 13
Sepsis (Infections and infestations) | 9 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Diphtheria (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pyrexia (General disorders) | 18 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Eyelid ptosis congenital (Congenital, familial and genetic disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Glomerulonephritis acute (Renal and urinary disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voxelotor (N=120) | Placebo (N=116)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 40 | 27
Anaemia (Blood and lymphatic system disorders) | 4 | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 2
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Pneumonia (Infections and infestations) | 1 | 1
Malaria (Infections and infestations) | 13 | 13
Upper respiratory tract infection (Infections and infestations) | 10 | 7
Tonsillitis (Infections and infestations) | 5 | 5
Bronchitis (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 4
Pharyngotonsillitis (Infections and infestations) | 3 | 3
Respiratory tract infection (Infections and infestations) | 3 | 6
Pharyngitis (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Varicella (Infections and infestations) | 2 | 2
Bacterial infection (Infections and infestations) | 1 | 1
Body tinea (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Mumps (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Carbuncle (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 4
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 15 | 10
Chest pain (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 1 | 3
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3
Blood bilirubin increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 2
Cardiac murmur (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Vitamin D decreased (Investigations) | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 3 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 4
Headache (Nervous system disorders) | 6 | 3
Dizziness (Nervous system disorders) | 1 | 2
Seizure (Nervous system disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Pallor (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 0 | 1
Night blindness (Eye disorders) | 1 | 0
Vernal keratoconjunctivitis (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Sickle cell nephropathy (Renal and urinary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Direct Billirubin (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT04218084/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT04218084/SAP_001.pdf